CLINICAL TRIAL: NCT04285658
Title: Pediatric KIDney Stone (PKIDS) Care Improvement Network
Acronym: PKIDS
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 19-016832; CER-2018C3-14778 (Other Grant/Funding Number: Patient-Centered Outcomes Research Institute)
Record Dates: First submitted 2020-02-24; First posted 2020-02-26 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Kidney Stone; Nephrolithiasis
Keywords: kidney; kidney stone; nephrolithiasis; Comparative Effectiveness; Patient Reported Outcomes
MeSH Terms: conditions — Kidney Calculi; Nephrolithiasis | interventions — Ureteroscopy; Nephrolithotomy, Percutaneous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Ureteroscopy
  Interventions: Procedure: Ureteroscopy
- Percutaneous Nephrolithotomy
  Interventions: Procedure: Percutaneous Nephrolithotomy
- Shock Wave Lithotripsy
  Interventions: Procedure: Shock Wave Lithotripsy

INTERVENTIONS:
Procedure: Ureteroscopy — An outpatient endoscopic surgery that accesses the ureters and kidneys per the urethra to fragment and remove the stones. Many patients who undergo ureteroscopy (URS), Shockwave lithotripsy (SWL), or percutaneous nephrolithotomy (PCNL) also have temporary tubes placed after the surgery to facilitate drainage, either internally (a stent) or externally (a nephrostomy tube).
  Other Names: URS
  Groups: Ureteroscopy
Procedure: Percutaneous Nephrolithotomy — A minimally invasive surgery in which a ~1cm flank incision is made, and a scope is passed through a tubular sheath into the kidney to fragment and remove the stone. There is typically a 1- to 2-day hospital stay. Many patients who undergo URS, SWL, or PCNL also have temporary tubes placed after the surgery to facilitate drainage, either internally (a stent) or externally (a nephrostomy tube).
  Other Names: PCNL
  Groups: Percutaneous Nephrolithotomy
Procedure: Shock Wave Lithotripsy — A non-invasive outpatient procedure that targets stones in the kidney or ureter with x-ray or ultrasound and uses shockwaves generated outside the body to fragment them; the fragments pass down the ureter and the patient expels them in the urine. Many patients who undergo URS, SWL, or PCNL also have temporary tubes placed after the surgery to facilitate drainage, either internally (a stent) or externally (a nephrostomy tube).
  Other Names: SWL
  Groups: Shock Wave Lithotripsy

SUMMARY:
The goals of this study are to improve the ability of pediatric patients and their caregivers to select surgical treatment options for kidney stones and to enable urologists to use techniques that result in the best outcomes for these surgeries.

DETAILED DESCRIPTION:
The rapid increase in the incidence of kidney stones among youth has resulted in a large population of patients who require surgery to removes stones but for whom little evidence exists to guide clinical care. Proper selection of surgical treatment options, which is directed by patient-specific factors and individual treatment goals, is the greatest determinant of successful outcomes.

This is a prospective cohort study. Investigators seek to compare stone clearance, re-treatment, and unplanned healthcare encounters for ureteroscopy, shockwave lithotripsy, and percutaneous nephrolithotomy.

Additionally, Investigators also seek to compare patients' experiences after ureteroscopy, shockwave lithotripsy, and percutaneous nephrolithotomy.

Setting/Participants:

This study will be conducted by the Pediatric KIDney Stone (PKIDS) Care Improvement Network, which includes 23 pediatric healthcare systems (25 sites) in the United States.

Patient participants include patients aged 8 to 21 years who undergo a surgical intervention for kidney stones as part of their clinical care. The surgical interventions include ureteroscopy, shockwave lithotripsy, and percutaneous nephrolithotomy, all of which would be performed as part of routine clinical care.

Study Interventions and Measures:

Stone clearance will be assessed with ultrasound (obtained as part of clinical care) 6 weeks after surgery, which is the standard of care at all PKIDS sites. Re-treatment and unplanned healthcare encounters will be assessed within the first 3 months after surgery. Patients' experiences will be measured through questionnaires administered pre-operatively and within 3 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, 8-21 years of age, undergoing planned URS, SWL, or PCNL for the removal of at least one kidney and/or ureteral stone.
2. Parental/guardian or participant (if ≥ 18 years old) permission (informed consent), and if appropriate, child assent

2a. Individuals who are not able to provide consent/assent (whether ≥18 or < 18 years) and/or not willing or able to complete questionnaires are eligible for participation for the stone clearance assessment and Electronic Health Record (EHR) surveillance if the legal guardian consents for study participation.

2b. Individuals for whom native-language questionnaires are not available can also participate in stone clearance assessment and EHR surveillance.

Exclusion Criteria:

1. Patients for whom conducting informed consent and baseline study procedures would confer additional risk (e.g. obstructing ureteral stone with fever requiring emergency surgery) and delay necessary immediate clinical care.
2. Parent/guardians or patients, who, in the opinion of the Investigator, may be non-compliant with study schedules or procedures

Ages: 8 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients in the United States receiving clinical care for kidney stones at a medical facility in the PKIDS Network.
Sampling Method: Non-Probability Sample
Enrollment: 1290 (Actual)
Dates: Start 2020-04-02 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Stone clearance | 6 weeks post-op +/- 2 weeks
  Presence or absence of kidney stones will be assessed via post-operative clinically-indicated renal bladder ultrasound.

SECONDARY OUTCOMES:
Patient-Reported Outcomes | Immediate impact (within 7 days) and delayed impact (up to 90 days) after surgery
  Patients' experiences before and after URS, SWL, and PCNL will be measured. Investigators will assess the immediate and delayed impact of surgery on patient-reported outcomes (PROs) selected by PKIDS patient partners. The patient reported outcomes (PROs) include the Patient-Reported Outcomes Measurement Information System (PROMIS), other questionnaires commonly used in studying the impact of kidney stone disease on health states, and urinary tract symptoms.
Patients' Experiences | Immediate impact (within 7 days) and delayed impact (up to 90 days) after surgery
  Investigators will examine Heterogeneity of Treatment Effect (HTE) by age and sex and identify modifiable surgical techniques that impact patient experiences for each surgery.
Patients' Experiences | Up to 90 days after surgery
  Investigators will also determine unplanned hospitalizations, emergency department (ED) visits, and repeat surgeries for the 3 months following each procedure to examine impact on patients' experiences.

CONTACTS AND LOCATIONS:
Locations (31):
- United States (30):
  - Children's of Alabama, Birmingham, Alabama
  - Children's Hospital Los Angeles, Los Angeles, California
  - UCLA Mattel Children's Hospital, Los Angeles, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Nemours A. I. duPont Hospital for Children, Wilmington, Delaware
  - Children's National Health System, Washington D.C., District of Columbia
  - University of Florida Health Shands Children's Hospital, Gainesville, Florida
  - Nemours Children's Specialty Care, Jacksonville, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Children's Hospital of Atlanta, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - University of Kentucky, Lexington, Kentucky
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - St. Louis Children's Hospital, St Louis, Missouri
  - Cohen Children's Medical Center, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Monroe Carell Jr. Children's Hospital at Vanderbilt, Nashville, Tennessee
  - Children's Medical Center of Dallas, Dallas, Texas
  - Texas Children's Hospital, Houston, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - Children's Hospital of Richmond at VCU, Richmond, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Children's Wisconsin, Milwaukee, Wisconsin
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tasian GE, Chu DI, Nelson CP, DeFoor WR, Ziemba JB, Huang J, Luan X, Kurtz M, Ching CB, Dangle P, Schaeffer AJ, Sturm R, Wu W, Bayne C, Fernandez N, Chua ME, DeMarco R, Ellsworth P, Augelli B, Bi-Karchin J, McCune RD, Vatsky S, Back S, Wang Z, Beck H, Kurth A, Kurth L, Pleskoff A, Forrest CB, Ellison JS; PKIDS Care Improvement Network; Rove K, Sparks S, Nelson E, Schlomer B, Krill A, Tong CMC, Taylor A, Ramachandra P, Stec A, Casale P, Coplen D, Janzen N, Bagley K, Denburg MR, Dickinson K, Laberee R, Lorenzo M, Selman-Fermin A, Dos Santos J, Grant C, Kraft K, Meenakshi-Sundaram B. Ureteroscopy vs Shockwave Lithotripsy to Remove Kidney Stones in Children and Adolescents: A Nonrandomized Clinical Trial. JAMA Netw Open. 2025 Aug 1;8(8):e2525789. doi: 10.1001/jamanetworkopen.2025.25789. PMID 40773197
- [Derived] Ellison JS, Lorenzo M, Beck H, Beck R, Chu DI, Forrest C, Huang J, Kratchman A, Kurth A, Kurth L, Kurtz M, Lendvay T, Sturm R, Tasian G; Pediatric KIDney Stone Care Improvement Network. Comparative effectiveness of paediatric kidney stone surgery (the PKIDS trial): study protocol for a patient-centred pragmatic clinical trial. BMJ Open. 2022 Apr 5;12(4):e056789. doi: 10.1136/bmjopen-2021-056789. PMID 35383073